CLINICAL TRIAL: NCT02771392
Title: Treatment of Corneal Abrasions With Topical Tetracaine: an Evaluation of Safety and Efficacy
Brief Title: Treatment of Corneal Abrasions With Topical Tetracaine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Charles Pereyra, Resident Physician, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA001
Record Dates: First submitted 2016-05-02; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Corneal Abrasion
MeSH Terms: conditions — Corneal Injuries | interventions — Saline Solution; Sodium Chloride; Solutions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetracaine Group (Experimental): Patients with he primary diagnosis of corneal abrasion will be treated with ophthalmic tetracaine. Tetracaine will be supplied in three plastic prefilled, commercially available vials, each containing 0.5 mL of preservative-free, undiluted 1% tetracaine hydrochloride (a total of 1.5 mL or approximately 50 drops will be provide to avoid overuse). Patients will be instructed to use 1-2 drops of up to every 30 min for pain control over a 48 hour period with subsequent followup with the ophthalmologist.
  Interventions: Drug: Ophthalmic Tetracaine
- Normal Saline Group (Placebo Comparator): Patients with the primary diagnosis of corneal abrasion will be treated with normal saline eye drops. Normal saline will be supplied in three plastic prefilled, commercially available vials, each containing 0.5 mL of normal saline. Patients will be instructed to use 1-2 drops of up to every 30 min for pain control over a 48 hour period with subsequent followup with the ophthalmologist.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ophthalmic Tetracaine — 1-2 drops to affected eye every 15-30 minutes over 24-48 hours as need
  Other Names: 1% tetracaine solution
  Arms: Tetracaine Group
Other: Normal Saline — 1-2 drops to affected eye every 15-30 minutes over 24-48 hours as need
  Other Names: sodium chloride in 0.85% solution
  Arms: Normal Saline Group

SUMMARY:
Corneal abrasion (CA) is one of the most common eye injuries, accounting for 10% of eye-related emergency visits.1 A 1985 survey showed that around 3% of all visits to US general practitioners were for corneal abrasions. In addition, in 2008, approximately 27,450 work-related eye injuries and illnesses occurred that caused missed time from work.1Due to the large number of nerve endings even small corneal injuries can produce significant pain. The discomfort is typically most pronounced in the first 24-48 hours, and in many cases showed a loss in time at work and disruption of daily activities. The current standard of care in the emergency department includes topical analgesia and antibiotics with a change to oral analgesics upon discharge. Despite the ineffectiveness of oral analgesics in treating CA pain, most physicians do not prescribe topical analgesics based on standard medical teaching. The study's aim is to further investigate the role of tetracaine in the outpatient management of CA utilizing models already established to ensure safety. To accomplish this investigators will employ a prospective, double blind, randomized control model to compare undiluted 1% tetracaine hydrochloride to normal saline in patients presenting to the ED with uncomplicated corneal abrasions. Tetracaine will be supplied in three plastic prefilled, commercially available vials, each containing 0.5 mL of preservative-free, undiluted 1% tetracaine hydrochloride (a total of 1.5 mL or approximately 50 drops will be provide to avoid overuse). Saline will also be supplied in three plastic prefilled, commercially available vials, plastic bullets. Follow up visits or calls will be provide at 48 hour to reevaluate symptoms an asses the patients perceived pain using VAS provided in participant introduction packet during the informed consent process.

DETAILED DESCRIPTION:
Corneal abrasion (CA) is one of the most common eye injuries, accounting for 10% of eye-related emergency visits.1 A 1985 survey showed that around 3% of all visits to US general practitioners were for corneal abrasions. In addition, in 2008, approximately 27,450 work-related eye injuries and illnesses occurred that caused missed time from work.1Due to the large number of nerve endings even small corneal injuries can produce significant pain. The discomfort is typically most pronounced in the first 24-48 hours, and in many cases showed a loss in time at work and disruption of daily activities. The current standard of care in the emergency department includes topical analgesia and antibiotics with a change to oral analgesics upon discharge. Despite the ineffectiveness of oral analgesics in treating CA pain, most physicians do not prescribe topical analgesics based on standard medical teaching. This teaching is extrapolated from data from case reports and animal studies reporting complications associated with long-term use; including addiction, infection, ulceration, and increased healing time. Previous studies have also rejected topical analgesia citing equivocal effectiveness and inconclusive safety data. However, all of the early human case reports described patients who used topical anesthetics inappropriately-either far too frequently, for too prolonged a treatment period, or with too concentrated an anesthetic. Contrary to the medical cannon, studies have now begun show the effectiveness of topical anesthetics in reducing pain, and safe application when given at low doses and when given in quantities lasting only 24-48 hours. A recent prospective, randomized trial, published in Academic Emergency Medicine, observed the efficacy and safety of tetracaine compared to normal saline in 116 patients presenting with uncomplicated CA. The intervention was either undiluted topical tetracaine hydrochloride 1% or saline, applied up to every 30 minutes for 24 hours. The study showed topical tetracaine used for 24 hours was safe, revealing no difference in complications between the two groups, with all individuals attaining full healing within 1 month. Additionally, median visual analog scale (VAS) pain scores were lower in the tetracaine group at all study time points after presentation, however statistical significance was not observed. Furthermore, patient surveys on overall effectiveness revealed that patients perceived tetracaine to be significantly more effective than saline. In fact, several researchers now recommend that the short-term use of tetracaine eye drops for 24 hours for pain relief from simple corneal abrasions should become routine practice. Nevertheless both skeptics and supporters agree that more research is needed in order to appropriately establish topical analgesics as a the standard of care. The importance of conducting research in the management of CA is underscored by the significant impact topical analgesics may provide in reliving patients pain compared to standard treatment. The study's aim is to further investigate the role of tetracaine in the outpatient management of CA utilizing models already established to ensure safety. This study will employ a prospective, double blind, randomized control model to compare undiluted 1% tetracaine hydrochloride to normal saline in patients presenting to the ED with uncomplicated corneal abrasions. Tetracaine will be supplied in three plastic prefilled, commercially available vials, each containing 0.5 mL of preservative-free, undiluted 1% tetracaine hydrochloride (a total of 1.5 mL or approximately 50 drops will be provide to avoid overuse). Saline will also be supplied in three plastic prefilled, commercially available vials, plastic bullets. Follow up visits or calls will be provide at 48 hour to reevaluate symptoms an asses the patients perceived pain using VAS provided in participant introduction packet during the informed consent process.

STUDY PROCEDURES

a. Study visits and parameters to be measured Patients will be assessed using a VAS upon follow up at 48 hours. Patients will also be evaluated for complications either by phone or at a follow-up visit, which is at the participants discretion. All patients will be encouraged to follow up with ophthalmology as-per standard protocol.

c. Drugs to be used (dose, method, schedule of administration, dose modifications, toxicities), include Toxicity Grading Scale (if applicable) Tetracaine will be supplied in three plastic prefilled, commercially available vials, each containing 0.5 mL of preservative-free, undiluted 1% tetracaine hydrochloride (a total of 1.5 mL or approximately 50 drops will be provide to avoid overuse). Patient will be instructed to use no more than 1-2 drops in the affected eye every 30 minutes while awake for 24-48 hours

STATISTICAL ANALYSIS

1. List of variables and their definition Variables will include perceived pain using a VAS, and overall perceived effectiveness of solution provided.
2. Outcome measures,endpoints The outcome of interest is weather-or-not tetracaine is superior to placebo in controlling pain caused by CA
3. Type of analysis A two sample T-test will be used comparing the average pain scale between the tetracaine and placebo group
4. Sample size of 100-200 patients is expected

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age with a primary diagnosis of uncomplicated corneal abrasion presenting to NYMH emergency department

Exclusion Criteria:

* Patients<18 years of age with complicated corneal abrasions or other eye injuries
* Present more than 36 hours after their initial injury
* Had previous eye surgery or cataracts
* Wear contact lenses or if their injury was caused from contact lens wear
* Had injured both eyes
* Unable to give informed consent
* Current infectious or chemical conjunctivitis
* Have a grossly contaminated foreign body in their eye
* Currently suffering from an ocular infection
* Currently or previously had herpes keratitis
* Allergies to tetracaine or similar medication classes
* Had an injury requiring urgent ophthalmologic evaluation; including penetrating eye injuries, large or complicated corneal abrasions, or injuries causing a significant disruption of visio)
* Unable to attend follow up in 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Pain assessed with Visual Analog Scale | Up to 24 months
  Participants receiving both arms of the study (Tetracaine and Normal Saline) will be provided with a Visual Analog Scale in there study welcome packet. Scales will be completed at the end of 48 hours and submitted at follow up visit or mailed in if visit is deferred.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Melville, M.D., Study Director — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data of pain perception and complications of patients

REFERENCES:
- [Background] Waldman N, Densie IK, Herbison P. Topical tetracaine used for 24 hours is safe and rated highly effective by patients for the treatment of pain caused by corneal abrasions: a double-blind, randomized clinical trial. Acad Emerg Med. 2014 Apr;21(4):374-82. doi: 10.1111/acem.12346. PMID 24730399
- [Background] Pruet CM, Feldman RM, Kim G. Re: "topical tetracaine used for 24 hours is safe and rated highly effective by patients for the treatment of pain caused by corneal abrasions: a double-blind, randomized clinical trial". Acad Emerg Med. 2014 Sep;21(9):1062-3. doi: 10.1111/acem.12470. No abstract available. PMID 25269590
- [Background] Swaminathan A, Otterness K, Milne K, Rezaie S. The Safety of Topical Anesthetics in the Treatment of Corneal Abrasions: A Review. J Emerg Med. 2015 Nov;49(5):810-5. doi: 10.1016/j.jemermed.2015.06.069. Epub 2015 Aug 15. PMID 26281814
- [Result] Segal KL, Fleischut PM, Kim C, Levine B, Faggiani SL, Banerjee S, Gadalla F, Lelli GJ Jr. Evaluation and treatment of perioperative corneal abrasions. J Ophthalmol. 2014;2014:901901. doi: 10.1155/2014/901901. Epub 2014 Feb 4. PMID 24672709
- [Derived] Algarni AM, Guyatt GH, Turner A, Alamri S. Antibiotic prophylaxis for corneal abrasion. Cochrane Database Syst Rev. 2022 May 27;5(5):CD014617. doi: 10.1002/14651858.CD014617.pub2. PMID 35622535